CLINICAL TRIAL: NCT03289650
Title: Once-Daily Extended-Release Tacrolimus vs. Twice-Daily Tacrolimus: Impact on T-Cell Subpopulations and Markers of Renal Tubule-toxicity in Kidney Transplant Patients
Brief Title: Extended Release Tacrolimus vs. Twice-Daily Tacrolimus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lorenzo Gallon (Other)
Responsible Party: Sponsor-Investigator, Lorenzo Gallon, Professor of Medicine, Northwestern University
Organization: Northwestern University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00205327
Record Dates: First submitted 2017-09-12; First posted 2017-09-21 (Actual); Results first posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: End Stage Renal Disease; Rejection of Renal Transplant
Keywords: immunosuppression
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of care tacrolimus twice-daily (Active Comparator)
  Interventions: Drug: Tacrolimus
- Extended-release tacrolimus once-daily (Active Comparator)
  Interventions: Drug: Tacrolimus Extended Release Oral Tablet [Envarsus]

INTERVENTIONS:
Drug: Tacrolimus — immunosuppressive agent tacrolimus, given twice-daily
  Arms: Standard of care tacrolimus twice-daily
Drug: Tacrolimus Extended Release Oral Tablet [Envarsus] — immunosuppressive agent extended-release tacrolimus, given once daily
  Other Names: LCP-tacro
  Arms: Extended-release tacrolimus once-daily

SUMMARY:
The overall aim of the study is to prospectively investigate the impact of two maintenance calcineurin inhibitor immunosuppressive regimens: once-daily extended release tacrolimus and twice-daily tacrolimus on subpopulations of T and B cells and alloreactive T cells as well as on renal allograft function.

DETAILED DESCRIPTION:
Kidney transplantation is the treatment of choice for most patients with end-stage renal disease. Lifelong immunosuppressive therapies are required to prevent organ rejection. However, long term exposure to immunosuppressive therapy after kidney transplantation can place patients at risk for multiple adverse events. The optimal immunosuppressive therapy is not well established. Tacrolimus, a calcineurin inhibitor (CNI) is highly effective in preventing acute rejection after organ transplantation (2). It is used as part of the immunosuppression regimen for the majority of kidney and liver transplant recipients (3). However, treatment with current formulation of Tacrolimus generates high peaks and low troughs in drug concentrations in the blood. It is known that high exposure to CNI is associated with renal toxicities and adverse events (4). New once-daily dosage formulations are now developed with the hope of minimizing side effects while maintaining excellent outcomes (5-8).

LCP-Tacro (Envarsus® XR, Veloxis Pharmaceuticals), a new once-daily formulation of tacrolimus, was approved by the FDA in 2015 for conversion from twice-daily tacrolimus in kidney transplant recipients. It is a prolonged-release tacrolimus formulation, utilizing a MeltDose drug delivery technology designed to improve the bioavailability of drugs with low water solubility (1). Recent clinical data demonstrated that once-daily LCP-Tacro has improved pharmacokinetic bioavailability, rapid achievement of therapeutic trough levels, less fluctuation and swing in whole blood concentration, non-inferior efficacy and similar safety, with lower tacrolimus dose than other tacrolimus formulations.

The target population is adult recipients of immediately functioning living and deceased donor renal allografts. Immediate function will be defined as the absence of the need for hemodialysis in the first week following renal transplantation.

Prospective randomized single center open label study of 2 groups of kidney transplant patients

* Group 1 : standard of care (SOC) control group will receive tacrolimus twice-daily (n=25)
* Group 2 : LCP-Tacro (Envarsus® XR) group will receive LCPT tablets once daily (n=25)

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are males or females aged 18-65 years. 2. Use of the following induction medications: basiliximab and rituximab. 2. Donors aged 18-65 years. 3. No prior organ transplant 4. Patients who are single-organ recipients (kidney only). 5. Women who are of childbearing potential must have a negative serum pregnancy test before transplantation and agree to use a medically acceptable method of contraception throughout the treatment period.

6. Subject (recipient) is able to understand the consent form and give written informed consent

Exclusion Criteria:

1. Delayed graft function (please see above).
2. Known sensitivity or contraindication to alemtuzumab, Envarsus® XR, tacrolimus or MMF.
3. Use of the following induction medications: basiliximab and rituximab
4. Patient with significant or active infection.
5. Patients with a positive flow cytometric crossmatch using donor lymphocytes and recipient serum.
6. Patients with PRA > 40%
7. Patients with current or historic donor specific antibodies
8. Body Mass Index (BMI) of < 18 or > 35
9. Patients who are pregnant or nursing mothers.
10. Patients whose life expectancy is severely limited by diseases other than renal disease.
11. Ongoing active substance abuse, drug or alcohol.
12. Major ongoing psychiatric illness or recent history of noncompliance.
13. Significant cardiovascular disease (e.g.):

    * Significant non-correctable coronary artery disease;
    * Ejection fraction below 30%;
    * History of recent myocardial infarction.
14. Malignancy within 3 years, excluding non-melanoma skin cancers.
15. Serologic evidence of infection with HIV or HBVs-Ag positive.
16. Patients with a screening/baseline total white blood cell count < 4,000/mm3; platelet count < 100,000/mm3; triglyceride > 400 mg/dl; total cholesterol > 300 mg/dl.
17. Investigational drug within 30 days prior to transplant surgery.
18. Anti-T cell therapy within 30 days prior to transplant surgery.
19. Diagnosis of atypical-Hemolytic Uremic Syndrome (aHUS).
20. Subjects transplanted with a Hepatitis C NAT-positive kidney.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Control Arm: Standard of Care (SOC) Tacrolimus: 1-2 mg 2x daily (BID), per SOC. The dose will be modified to achieve 12 hours trough concentrations of 8-12 ng/ml
- Group 2: Interventional Arm: Study Related Drug: LCP-Tacrolimus/Envarsus XR (LCP-Tacro/Envarsus XR): One 5mg extended-release tablet taken once daily (QD) to achieve a 24-hour trough concentrations of 8-12 ng/ml
Period: Overall Study
Arm/Group | Group 1: Control Arm: Standard of Care (SOC) Tacrolimus | Group 2: Interventional Arm: Study Related Drug: LCP-Tacrolimus/Envarsus XR (LCP-Tacro/Envarsus XR)
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Tacrolimus Twice-daily | Extended-release Tacrolimus Once-daily | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.14 (12.7) | 47.53 (16.04) | 45.4 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 10 | 13 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Cause of Kidney Disease [Number; unit: participants]
  Diabetes | 3 | 4 | 7
  Glomerulonephritis | 3 | 4 | 7
  Obstructive Nephropathy | 2 | 0 | 2
  Congenital | 1 | 2 | 3
  Others | 5 | 5 | 10
Type of Donor [Count of Participants; unit: Participants]
  Cadaveric | 0 | 1 | 1
  Living | 14 | 14 | 28
Panel reactive antibodies (PRA) [Mean (Standard Deviation); unit: percentage]
  Major histocompatibility complex class I (MHC-I) antibodies | 1.93 (2.79) | 4.20 (8.44) | 3.1 (6.4)
  Major histocompatibility complex class II (MHC-II) antibodies | 3.07 (5.18) | 4.07 (9.01) | 3.6 (7.3)
Estimated glomerular filtration rate (eGFR) [Median (Standard Deviation); unit: ml/min/1.73m2] — measured in mL/min/1.73m^2. MDRD equation was used to calculate GFR, using age, sex, race and serum creatinine
  ml/min/1.73m2 | 52.43 (9.26) | 51.77 (9.69) | 52.1 (10.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Kidney Transplant Function From 2 Weeks Post Transplant Through 12 Months Post Transplant
Description: change in the mean eGFR from the baseline (2 weeks post transplant), 3 months (post transplant) , and 12 months (post transplant).
Time Frame: 2 weeks post transplant through 12 months post transplant
Measure: Mean (Standard Error); unit: mL/min/1.73m^2
Groups:
- Group 1: Control Arm: Standard of Care (SOC) Tacrolimus: Tacrolimus: immunosuppressive agent tacrolimus, 1-2 mg 2x daily (BID), per SOC. The dose will be modified to achieve 12 hours trough concentrations of 8-12 ng/ml
- Group 2: Interventional Arm: Study Related Drug: LCP-Tacrolimus/Envarsus XR (LCP-Tacro/Envarsus XR): Tacrolimus Extended Release Oral Tablet [Envarsus]: immunosuppressive agent extended-release tacrolimus, One 5mg extended-release tablet taken once daily (QD) to achieve a 24-hour trough concentrations of 8-12 ng/ml
Arm/Group | Group 1: Control Arm: Standard of Care (SOC) Tacrolimus | Group 2: Interventional Arm: Study Related Drug: LCP-Tacrolimus/Envarsus XR (LCP-Tacro/Envarsus XR)
Number analyzed (Participants) | 14 | 15
mL/min/1.73m^2 | 2.03 (1.71) | -2.19 (1.77)

2. Secondary Outcome: Change in Subpopulations of T Cells From 2 Weeks Post Transplant Through 12 Months Post Transplant
Description: Blood, urine and kidney tissue analysis via serial flow cytometric immunophenotyping (includes regulatory T and B cell populations as well as immune functions).
Time Frame: Measured at 2 weeks post transplant, 3 months post transplant, 12 months post transplant
Population: Secondary outcome data will not be reported because support to collect secondary data was not present
Arm/Group | Group 1: Control Arm: Standard of Care (SOC) Tacrolimus | Group 2: Interventional Arm: Study Related Drug: LCP-Tacrolimus/Envarsus XR (LCP-Tacro/Envarsus XR)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Acute Rejection at 3 Months and 12 Months Post-Transplant
Description: Acute rejection of kidney transplant is determined via biopsy.
Time Frame: Measured at 3 months post transplant, 12 months post transplant
Measure: Count of Participants; unit: Participants
Groups:
- Group 2: Interventional Arm: Study Related Drug: LCP-Tacrolimus/Envarsus® XR (LCP-Tacro/Envarsus XR): One 5mg extended-release tablet taken once daily (QD) to achieve a 24-hour trough concentrations of 8-12 ng/ml
Arm/Group | Group 1: Control Arm: Standard of Care (SOC) Tacrolimus | Group 2: Interventional Arm: Study Related Drug: LCP-Tacrolimus/Envarsus® XR (LCP-Tacro/Envarsus XR)
Number analyzed (Participants) | 14 | 15
Participants
  Acute rejection at 3 months | 0 | 1
  Acute rejection at 12 months | 0 | 2

4. Secondary Outcome: Number of Participants With Graft Loss at 3 Months and 12 Months Post-Transplant
Description: Graft loss is determined via biopsy.
Time Frame: Measured at 3 months post transplant, 12 months post transplant
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Control Arm: Standard of Care (SOC) Tacrolimus: Tacrolimus: immunosuppressive agent Tacrolimus 1-2 mg 2x daily (BID), per SOC. The dose will be modified to achieve 12 hours trough concentrations of 8-12 ng/ml-daily
Arm/Group | Group 1: Control Arm: Standard of Care (SOC) Tacrolimus | Group 2: Interventional Arm: Study Related Drug: LCP-Tacrolimus/Envarsus XR (LCP-Tacro/Envarsus XR)
Number analyzed (Participants) | 14 | 15
Participants
  Graft Loss at 3 months | 0 | 0
  Graft loss at 12 months | 0 | 0

5. Secondary Outcome: Number of Subjects Deceased at at 3 Months and 12 Months Post-Transplant
Description: Subject survival status is continually monitored via routine follow-up visits.
Time Frame: Through 12 months post transplant
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Control Arm: Standard of Care (SOC) Tacrolimus: Tacrolimus: immunosuppressive agent Tacrolimus 1-2 mg 2x daily (BID), per SOC. The dose will be modified to achieve 12 hours trough concentrations of 8-12 ng/ml
- Group 2: Interventional Arm: Study Related Drug: LCP-Tacrolimus/Envarsus® XR (LCP-Tacro/Envarsus XR): Tacrolimus Extended Release Oral Tablet [Envarsus]: immunosuppressive agent extended-release One 5mg extended-release tablet taken once daily (QD) to achieve a 24-hour trough concentrations of 8-12 ng/ml
Arm/Group | Group 1: Control Arm: Standard of Care (SOC) Tacrolimus | Group 2: Interventional Arm: Study Related Drug: LCP-Tacrolimus/Envarsus® XR (LCP-Tacro/Envarsus XR)
Number analyzed (Participants) | 14 | 15
Participants
  Subject Death at 3 months | 0 | 0
  Subject Death at 12 months | 0 | 0

6. Secondary Outcome: Number of Participants With Change in Allograft Immunohistopathology Profile
Description: Tissue analysis via immunohistopathological staining and microscopic examination Moderate acute tubular necrosis => presence of focal coagulative necrosis or infarction on histopathologic examination
  Arteriolar hyalinosis grade 2 means: Replacement of degenerated smooth muscle cells by hyaline deposits in more than 1 arteriole, without circumferential involvement
  Global glomerulosclerosis >grade 2, means glomerulosclerosis affecting more than 50% of glomeruli in the biopsy sample
  IFTA : Interstitial fibrosis and tubular atrophy: Inflammation in 26% to 50% of scarred cortical parenchyma
Time Frame: Measured at 3 months post transplant, 12 months post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Control Arm: Standard of Care (SOC) Tacrolimus | Group 2: Interventional Arm: Study Related Drug: LCP-Tacrolimus/Envarsus XR (LCP-Tacro/Envarsus XR)
Number analyzed (Participants) | 14 | 15
Participants
  Acute tubular necrosis > moderate >=2 | 2 | 2
  Arteriolar Hyalinosis >= grade 2 | 2 | 2
  isometric vacuolization of tubules | 0 | 1
  Arteriolar myocyte vacuolization | 0 | 0
  Thrombotic microangiopathy | 1 | 1
  Global glomerulosclerosis >grade 2 | 1 | 2
  IFTA > grade 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were reviewed at 1 year after tranplant
Arm/Group | Standard of Care Tacrolimus Twice-daily | Extended-release Tacrolimus Once-daily
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/15
Other Adverse Events (participants affected / at risk) | 7/14 | 5/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Tacrolimus Twice-daily (N=14) | Extended-release Tacrolimus Once-daily (N=15)
Hospitalizations (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Tacrolimus Twice-daily (N=14) | Extended-release Tacrolimus Once-daily (N=15)
Infections (Immune system disorders) | 1 (1) | 1 (1)
Malignancy (Immune system disorders) | 0 (0) | 0 (0)
Leukopenia (Immune system disorders) | 4 (4) | 4 (4)
BK Viremia (Renal and urinary disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The study ran out of funding and as a result the outcome (Change in Subpopulations of T Cells) has not been analyzed. The PI will look for additional funding to complete the analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT03289650/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT03289650/ICF_001.pdf